CLINICAL TRIAL: NCT02922920
Title: Effects of Tart Cherry Juice on the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Sheau Ching Chai, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15A00149
Record Dates: First submitted 2016-09-20; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Risk Factors; Age-Related Cognitive Decline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tart cherry juice (Experimental): Participants consumed 16 fl. oz of tart cherry juice daily for 12 weeks.
  Interventions: Other: Tart cherry juice
- Placebo juice (Placebo Comparator): Participants consumed 16 fl. oz of placebo daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Tart cherry juice — 16 fl. oz of tart cherry juice
  Arms: Tart cherry juice
Other: Placebo — 16 fl. oz of placebo
  Arms: Placebo juice

SUMMARY:
Tart cherries are a rich source of antioxidants. Studies have shown that tart cherries exert anti-oxidative and anti-inflammatory properties. The purpose of this study is to learn about the effects of drinking tart cherry juice on cardiovascular and cognitive health.

DETAILED DESCRIPTION:
Thirty-seven older adults were randomly assigned to drink 16 oz per day of either tart cherry juice or placebo drink for 12 weeks. Blood and urine samples were collected at baseline and 12 weeks to assess biomarkers. Physical activity and 3-day diet records were also collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

• Age 65-80

Exclusion Criteria:

* Allergic to tart cherries
* Heavy smoker
* Taking medications that affect cognitive function
* History of neurological disorders
* History of traumatic brain injury
* History of stroke
* Clinical diagnosis of diabetes
* Clinical diagnosis of Alzheimer's Disease/Dementia
* GI disease
* Kidney disease
* Liver disease
* Cancer

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Baseline and 12 weeks
  Change from baseline in cognitive test performance at 12 weeks

SECONDARY OUTCOMES:
Cardiovascular risk factors | Baseline and 12 weeks
  Fasting blood samples were collected at baseline and 12 weeks. Change from baseline in cardiovascular risk factors including blood lipid profiles, atherogenic risk ratios, blood glucose, hemoglobin A1c, insulin, and blood pressure at 12 weeks.
Oxidative stress markers | Baseline and 12 weeks
  Fasting blood samples were collected at baseline and 12 weeks. Change from baseline in plasma 8-oxoguanine (ng/ml), plasma 8-hydroxy-2deoxy-guanosine (ng/mL), plasma hydroxynonenal (ng/ml), and plasma malondialdehyde (pmole/L) at 12 weeks.
Inflammatory markers | Baseline and 12 weeks
  Fasting blood samples were collected at baseline and 12 weeks. Change from baseline in plasma tumor-necrosis factor-α (pg/mL) and plasma high-sensitivity C-reactive protein (ng/mL) at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sheau Ching Chai, PhD, RD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No